CLINICAL TRIAL: NCT07242235
Title: Immediate Effects of Transcutaneous Electrical Nerve Stimulation on the Lumbar Erector Spinae Muscles' Stiffness and Pain: A Randomized Controlled Trial
Brief Title: Immediate Effects of TENS on Lumbar Erector Spinae Stiffness in Low Back Pain
Acronym: TENS-LUMBAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Amasya University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Dr., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETU-TENS-LBP-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Non-specific Low Back Pain; Lumbar Muscle Stiffness
Keywords: TENS; Low Back Pain; Muscle Stiffness; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) to active TENS or control/rest; both groups are assessed pre- and immediately post-intervention
Who Masked: Outcomes Assessor
Masking Description: The assessor who performs Myoton and VAS measurements will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: TENS (Experimental): Participants receive a single 30-minute session of conventional TENS applied bilaterally over the lumbar paraspinal (erector spinae) region. Pre- and post-intervention Myoton and VAS measurements are taken.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Control: Rest/Positioning (Other): Participants are positioned in the same way and remain at rest for 20 minutes without active TENS. Pre- and post-intervention Myoton and VAS measurements are taken.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Conventional TENS; frequency 80-100 Hz, pulse width 100-150 μs, intensity adjusted to strong but comfortable sensory level without muscle contraction; total duration 20 minutes; electrodes placed bilaterally at lumbar erector spinae level.
  Other Names: Rest/Observation

SUMMARY:
Low back pain is frequently associated with increased tone and stiffness of the lumbar erector spinae muscles, which may contribute to pain and functional limitation. Transcutaneous electrical nerve stimulation (TENS) is a non-invasive, safe, and widely used modality for pain reduction, but its very short-term (immediate) effects on lumbar muscle stiffness have not been clearly demonstrated. This randomized controlled trial will compare a single 20-minute session of conventional TENS with a control/rest condition in patients with non-specific low back pain. The primary outcomes will be change in lumbar erector spinae muscle stiffness (Myoton) and change in pain intensity (VAS) from baseline to immediately after the intervention. We hypothesize that TENS will produce a greater immediate reduction in muscle stiffness and pain than control.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal problems and often presents with increased paraspinal muscle activity and perceived stiffness around the lumbar region. Increased stiffness of the lumbar erector spinae may perpetuate pain and restrict movement. TENS provides afferent stimulation that can modulate pain through gate-control and descending inhibitory mechanisms and may secondarily reduce muscle tone. However, evidence about its acute influence on objective muscle stiffness parameters in LBP is limited.

This single-center, parallel-group, randomized controlled trial will recruit adults with chronic or recurrent non-specific low back pain who meet the eligibility criteria. Participants will be randomly assigned (1:1) to (1) an experimental group receiving conventional TENS applied bilaterally over the lumbar paraspinal area for 20 minutes (frequency ~80-100 Hz, pulse width ~100-150 μs), or (2) a control group undergoing the same positioning and timing without active TENS. All assessments will be performed immediately before and immediately after the intervention by an outcome assessor blinded to group allocation.

Primary outcomes are: (a) lumbar erector spinae muscle stiffness measured with a handheld myotonometer (e.g. Myoton) at standardized lumbar levels, and (b) pain intensity measured with a 10-cm visual analog scale (VAS). Secondary observations may include participant-reported comfort/tolerance of TENS and adverse events. The study is designed as a short-term physiological and symptomatic trial; no long-term follow-up is planned. Ethical approval was obtained from the Erzurum Technical University Ethics Committee (Meeting 13, Decision 04, 18.09.2025)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years

Non-specific low back pain persisting or recurring for ≥3 months

Reported tenderness/stiffness on palpation of the lumbar erector spinae muscles

Able to understand the study procedures and provide written informed consent

Able to attend on the same day for TENS application and pre-/post-intervention measurements

Exclusion Criteria:

* Low back pain with a specific cause (e.g. lumbar disc herniation with radiculopathy, infection, tumor, fracture, severe deformity)

Open wound, dermatitis, or any skin condition in the lumbar area that prevents electrode placement

Presence of a cardiac pacemaker or other implanted electronic device

Electrotherapy, injection, or manual therapy applied to the lumbar region within the previous 48 hours

Pregnancy

Severe neurological deficit or sensory loss

Use of analgesics/NSAIDs at a level that may interfere with pain or stiffness assessment at the time of evaluation

Any other condition deemed unsafe or inappropriate by the investigator

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in lumbar erector spinae muscle stiffness | Baseline (pre-intervention) and immediately post-intervention (within ~5 minutes of completing the 20-minute session)
  Muscle stiffness of the lumbar erector spinae will be measured with a handheld myotonometer (e.g. Myoton) at standardized lumbar levels. The outcome is the change score (post - pre) between TENS and control groups. Lower values indicate reduced stiffness.
Change in pain intensity (VAS) | Baseline (pre-intervention) and immediately post-intervention (within ~5 minutes of completing the 20-minute session)
  Pain intensity will be assessed using a 10-cm Visual Analog Scale (0 = no pain, 10 = worst pain). The outcome is the change score (post - pre) to compare TENS and control groups. Lower scores indicate pain reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan YAĞIZ, Dr., Principal Investigator — Amasya University
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is small, single-center, and includes identifiable clinical measurements that could risk participant privacy despite de-identification.